CLINICAL TRIAL: NCT01455493
Title: A Multicenter, Single-Arm, Open-Label, Phase II Study of GDC-0980 for The Treatment of Recurrent or Persistent Endometrial Carcinoma
Brief Title: A Study of GDC-0980 in the Treatment of Recurrent or Persistent Endometrial Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PIM4972g
Record Dates: First submitted 2011-10-18; First posted 2011-10-20 (Estimated); Last update posted 2016-08-11 (Estimated); Status verified 2016-08

CONDITIONS: Endometrial Carcinoma
MeSH Terms: conditions — Endometrial Neoplasms | interventions — 1-(4-((2-(2-aminopyrimidin-5-yl)-7-methyl-4-morpholinothieno(3,2-d)pyrimidin-6-yl)methyl)piperazin-1-yl)-2-hydroxypropan-1-one

ARMS (1):
- A (Experimental)
  Interventions: Drug: GDC-0980

INTERVENTIONS:
Drug: GDC-0980 — Oral daily dose

SUMMARY:
This is a multicenter, single-arm, open-label Phase II study to evaluate the activity of GDC-0980 in patients with recurrent or persistent endometrial cancer. The safety, tolerability, and pharmacokinetics of GDC-0980 will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have recurrent or persistent endometrial carcinoma that is refractory to curative therapy or established treatments
* Histologic confirmation of the original primary tumor is required
* Histologic or cytologic confirmation of the recurrent/progressive disease is desired
* Patients must have had at least one but no more than two prior chemotherapeutic regimens for management of endometrial carcinoma
* Disease that is measurable per RECIST v1.1
* No active infection requiring antibiotics
* Any hormonal therapy directed at the malignant tumor must be discontinued at least 2 weeks prior to first study treatment
* Any other prior therapy directed at the malignant tumor, including immunologic agents and radiotherapy, must be discontinued at least 2 weeks prior to first study treatment
* Adequate hematologic and end organ function

Exclusion Criteria:

* Type I diabetes or Type II diabetes requiring insulin
* Prior use of mTOR/PI3K inhibitor
* Current dyspnea at rest or any requirement for supplemental oxygen therapy to perform activities of daily living
* Previous diagnosis of pulmonary fibrosis of any cause
* History of myocardial infarction or unstable angina within 6 months prior to first study treatment
* Congestive heart failure
* History of malabsorption syndrome or other condition that would interfere with enteral absorption
* Clinically significant history of liver disease, including cirrhosis and current alcohol abuse
* Presence of positive test results for hepatitis B or hepatitis C
* Known HIV infection
* Active autoimmune disease that is not controlled by nonsteroidal anti inflammatory drugs
* Need for current chronic corticosteroid therapy
* Pregnancy, lactation, or breastfeeding
* Current severe, uncontrolled systemic disease
* Major surgical procedure or significant traumatic injury within 28 days prior to Day 1 or anticipation of the need for major surgery during the course of study treatment
* Uncontrolled hypercalcemia
* Leptomeningeal disease as a manifestation of cancer
* Known untreated or active brain metastases
* Grade >=2 hypercholesterolemia or hypertriglyceridemia

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2011-12; Primary Completion 2013-03 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Objective tumor response as assessed by the investigator using RECIST v1.1 | up to approximately 23 months
Progression-free survival (PFS), defined as the time from the first GDC-0980 treatment to disease progression as assessed by the investigator using RECIST v1.1, or death from any cause while on study | at 6 months

SECONDARY OUTCOMES:
Overall survival (OS), defined as the time from treatment initiation until death from any cause | up to approximately 36 months
Duration of objective tumor response defined as the time from first observation of an objective tumor response until first observation of disease progression as assessed by the investigator using RECIST v1.1 | up to approximately 23 months
Incidence of adverse events | up to approximately 23 months
Nature of adverse events | up to approximately 23 months
Severity of adverse events | up to approximately 23 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Genentech, Inc.
Locations (26):
- United States (26):
  - Phoenix, Arizona
  - Newport Beach, California
  - Orange, California
  - Palo Alto, California
  - San Francisco, California
  - Denver, Colorado
  - New Haven, Connecticut
  - Boca Raton, Florida
  - Orlando, Florida
  - West Palm Beach, Florida
  - Hinsdale, Illinois
  - Indianapolis, Indiana
  - Louisville, Kentucky
  - Scarborough, Maine
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Voorhees Township, New Jersey
  - New York, New York
  - Durham, North Carolina
  - Winston-Salem, North Carolina
  - Oklahoma City, Oklahoma
  - Abington, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Salt Lake City, Utah
  - Seattle, Washington
  - Milwaukee, Wisconsin